CLINICAL TRIAL: NCT04858542
Title: Developing Educational Modules to Improve Communication and Vocal Health Among Mask-wearing Healthcare Workers: Phase 2 of the COVID-19 Critical Community Challenge Grant
Brief Title: Evaluating the Impact of Vocal Health Education on Mask-wearing Workers During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Victoria McKenna, Assistant Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-0889
Record Dates: First submitted 2021-03-22; First posted 2021-04-26 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Health Behavior
Keywords: voice; communication
MeSH Terms: conditions — Health Behavior; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mask-wearing healthcare workers (Experimental): All participants in this arm will view the educational health modules and their subjective/objective outcomes will be measure pre/post module viewing.
  Interventions: Behavioral: Educational Vocal Health Modules

INTERVENTIONS:
Behavioral: Educational Vocal Health Modules — We have developed four educational health modules (total duration of approximately 30 minutes). First, these modules explain how masks impact communication and voice, then they describe health strategies to improve communication and voice, and finally, they give real-life examples of how the strategies can be implemented into the work setting.

SUMMARY:
The purpose of this clinical trial is to understand how viewing educational health modules impacts vocal health behaviors in mask-wearing healthcare workers.

DETAILED DESCRIPTION:
Results of the investigators' previous work showed that mask-wearing healthcare workers have difficulty with voice and communication. Healthcare workers reported significant increases in vocal effort and dyspnea while wearing masks, and showed greater effort and poorer vocal quality at the end of the workday compared to the beginning of the day. Despite these negative changes, very few healthcare workers reported using any type of communication strategy (e.g., taking breaks, using gestures). Therefore, the investigators developed educational modules to address the voice and communication problems facing this population. This clinical trial plans to evaluate how these educational modules impact subjective/objective voice and communication measures in mask-wearing healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* English Speaker
* Occupational voice user who is required to wear a mask at work

Exclusion Criteria:

* History of neurological disorder or disease
* History of head/neck cancer
* Current speech, language, voice, or hearing problem/disorder
* Currently sick or have been sick within the last 14 days, or is waiting on a COVID-19 test result

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in amount of Vocal Effort after 1 week | Assessed prior to module viewing and again 1-week later
  A self-perceptual rating of voice exertion and how hard it is to make a voice. The vocal effort scale will be rated on a 100-mm visual analog scale in which the left side (score of 0) indicates "no effort" to produce a voice, and the right side (score of 100) indicates "the most effort" to create a voice.
Learning of Health Information | Assessed immediately after viewing the modules
  Answer questions about the content of the module (short answer, multiple choice, true/false)

SECONDARY OUTCOMES:
Change in Relative fundamental frequency | Assessed prior to viewing modules, and then 1-week later
  An acoustic measure that characterizes change in fundamental frequency during voicing transitions. Participants will complete vowel-voiceless consonant-vowel combinations (e.g., /ifi/) and relative fundamental frequency will be determined.
Module Information Retention | Assessed at second session
  Answer question about the content of the modules (short answer, multiple choice, true/false)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria McKenna, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- Victoria McKenna, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lab website with contact information — https://vsmechlab.com